CLINICAL TRIAL: NCT01386216
Title: Phase I, Non-Randomized, Feasibility Study for the Use of Bone Marrow Cell Concentrate Prepared Using the Magellan System for the Treatment of Critical Limb Ischemia
Brief Title: Safety Study of Bone Marrow Cell Concentrate Prepared Using the Magellan System to Treat Critical Limb Ischemia (CLI)
Acronym: CLI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arteriocyte, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ART 10-001
Record Dates: First submitted 2011-06-29; First posted 2011-07-01 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Critical Limb Ischemia (CLI); Peripheral Vascular Disease (PVD)
Keywords: Critical limb ischemia; Peripheral vascular disease; platelet-rich plasma
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bone Marrow Cell Concentrate (Experimental): Bone Marrow Cell Concentrate Prepared Using the Magellan System
  Interventions: Device: Magellan®

INTERVENTIONS:
Device: Magellan® — Autologous Bone Marrow Cell Concentrate Prepared Using the Magellan System to be injected into the ischemic muscle tissue at 0.5 cc/injection for a total of 12-20 cc.
  Other Names: autologous cell concentrate

SUMMARY:
The purpose of this study is to evaluate the safety of administration of marrow-derived autologous hematopoietic stem cells (HSC) concentrate and platelet-rich plasma (PRP) gel for the treatment of Critical Limb Ischemia (CLI).

DETAILED DESCRIPTION:
Critical limb ischemia (CLI) continues to be an important cause of atherosclerotic morbidity and mortality despite conventional therapies. Modulation of angiogenesis is a promising alternative to surgical revascularization. Trials of isolated angiogenic growth factor therapies using recombinant proteins or gene transfer have been conducted, but with disappointing results because it is unlikely that a single angiogenic factor is solely or even primarily responsible for angiogenesis. Emerging stem cell therapies represent a new approach to the modulation of angiogenesis. Pluripotent hematopoietic stem cells (HSC) hold promise because they can reproduce a pro-angiogenic milieu in the ischemic limb rather than upregulate a single angiogenic factor.

For this CLI study, the Magellan® System is utilized for the preparation of autologous cell concentrate at the point of care. The bone marrow aspirate is obtained from the patient and concentrated with the cell concentration kit, and delivered intramuscularly to the affected limb for the treatment of impaired ischemic tissue in order to improve perfusion, reduce pain and revascularize tissues in patients who have inadequate tissue blood flow, prohibitive medical comorbidities, or failed previous treatments for revascularization for the prevention of amputation.

ELIGIBILITY:
Inclusion Criteria:

* Is able to provide written informed consent prior to study entry
* Is male or female, 18 - 85 years of age
* CLI with rest pain, tissue loss, or gangrene
* No option for revascularization as a result of one of the following:

  * failed previous revascularization, such as recurrent instant restenosis or graft occlusion.
  * inadequate target vessels as determined by baseline CTA/angiogram at the time of enrollment.
  * or prohibitive medical comorbidities such as high risk cardiovascular or pulmonary disease which would restrict operative procedures
  * Final determination of no option for revascularization will be made by a vascular surgeon not associated with the clinical trial.
* ABI less than 0.7, ankle pressure < 50 mmHg, or toe pressure < 30 mmHg.
* TcPO2 < 40 mmHg
* SPP < 35 mmHg
* Female subjects must be of non childbearing potential (defined as postmenopausal for at least 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy or hysterectomy]) or must be using adequate contraception (practicing one of the following methods of birth control):

  * Total abstinence from sexual intercourse (minimum of one complete menstrual cycle before study entry),
  * A partner who is physically unable to impregnate the subject (e.g., vasectomized)
  * Contraceptives (oral, parenteral, or transdermal) for 3 consecutive months prior to patient's cell concentrate administration,
  * Intrauterine device (IUD), or
  * Double barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream)
* If female is of childbearing potential, subject must have a negative serum pregnancy test at screening
* Confirmation of age-appropriate cancer screening consistent with the American Cancer Society guidelines

Exclusion Criteria:

* Patients with vascular lesions amenable to percutaneous intervention or where surgical bypass is indicated.
* Any contraindication to stem cell or platelet-rich plasma therapy.
* Isolated aorto-iliac stenoses or occlusions without infra-inguinal disease.
* Pregnancy
* Hemoglobin A1c >10 % on day of enrollment.
* Have an active malignancy or have undergone treatment for a malignancy in the preceding 5 years, with the exception of successful treatment of non-melanoma skin cancer.
* Stage 4 or greater chronic kidney disease (eGFR < 30 ml/min, MDRD estimate)
* Hemoglobin < 10 g/dl.
* Thrombocytopenia < 100,000 platelets/µL.
* Unwilling or unable to comply with follow-up visits.
* Proliferative retinopathy as determined by baseline retinal exam.
* Is unable to refrain from nicotine, caffeine and alcohol for a period beginning 24 hours prior to the treatment visit
* Has received an investigational medication or other study trial participation within 30 days prior to the Treatment Visit

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-04; Primary Completion 2016-04 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure or death | Baseline - 12 months
  Treatment failure is defined as major amputation

SECONDARY OUTCOMES:
Perfusion and Quality of Life measurements | Baseline - 12 months
  * Perfusion rate in treated tissue by measure of ankle-brachial index (ABI)
  * Perfusion rate in treated tissue by transcutaneous PO2 (TcPO2)
  * Perfusion rate in treated tissue by skin perfusion pressure (SPP)
  * Pain intensity using Visual Analogue Scale (VAS)
  * Quality of Life (QoL) by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michael Go, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States